CLINICAL TRIAL: NCT04121819
Title: Cytarabine Monotherapy for Adult Patients With Newly Diagnosed Langerhans Cell Histiocytosis: A Single Arm, Single Center, Prospective Phase 2 Study
Brief Title: AraC for Newly Diagnosed Adult Langerhans Cell Histiocytosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Cao Xinxin, Associate Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCHNDLCH2
Record Dates: First submitted 2019-10-07; First posted 2019-10-10 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Langerhans Cell Histiocytosis
Keywords: Langerhans cell histiocytosis; adult; newly diagnosed
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — Cytarabine

STUDY DESIGN:
Intervention Model Description: AraC
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AraC (Experimental): cytarabine 100mg/m2 d1-5 subcutaneous
  Interventions: Drug: Cytarabine

INTERVENTIONS:
Drug: Cytarabine — cytarabine 100mg/m2 d1-5 subcutaneous

SUMMARY:
Langerhans cell histiocytosis (LCH) is a rare, heterogeneous histiocytic disorder occurring in patients of all ages from neonates to the elderly. The current standard treatment protocol for children with de novo multisystem LCH is vinblastine plus prednisone. This regimen has never been proven effective for adults in a prospective study, since the only prospective trial evaluating the efficacy of a vinblastine/prednisone regimen in adults was prematurely closed due to unacceptable toxicities. A retrospective study showed an advantage for cytarabine monotherapy compared with vinblastine/prednisone in bone LCH patients. This phase 2, prospective, single-center study is designed to evaluate the efficacy and safety of cytarabine monotherapy in adults with newly diagnosed MS-LCH or LCH with multifocal single system (SS-m) involvement.

ELIGIBILITY:
Inclusion Criteria:

* • Histologically confirmed diagnosis of LCH.

  * Patients were newly diagnosed or did not receive prior systemic treatment of LCH (patients who had received radiotherapy alone were allowed).
  * Age ≥18 years and ≤75 years.
  * LCH involved multisystem or multifocal single system.
  * Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
  * Patients must have adequate renal, liver, and bone marrow function as defined by the following criteria:

    * Absolute neutrophil count ≥1500 cells per mm3 or ≥500 cells per mm3 in the case of known hematopoietic system involvement by LCH.
    * Platelet count ≥100000 cells per mm3 or ≥20000 cells per mm3 in the case of known hematopoietic system involvement by LCH.
    * Creatinine clearance [according to Cockcroft formula] ≥60 mL/min.
    * Aspartate aminotransferase and alanine aminotransferase ≤2·5×upper limit of normal [ULN], and total bilirubin ≤2·5×ULN; or ≤10×ULN in the case of known liver involvement by LCH.
  * No active or untreated infection.
  * No cardiac abnormalities.
  * Subject provide written informed consent.
  * A female is eligible to enter and participate in this study if she is of:

    * Non-childbearing potential including ω Any female who has had a surgical procedure rendering her incapable of becoming pregnant.

ω Subjects have experienced total cessation of menses for more than 1 year and be greater than 45 years in age.

⎫ Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, and agrees to use adequate contraception.

Male subjects must use an effective barrier method of contraception during the study and for 90 days following the last course of MA if sexually active with a childbearing potential

Exclusion Criteria:

* • Non-langerhans cell histiocytosis.

  * Patients had concurrent malignancies.
  * Patients who had received any treatment except radiotherapy for LCH.
  * History of myocardial infarction, or unstable angina, or New York Heart Association (NYHA) Grade III-IV within 6 months prior to Day 1.
  * Women who were pregnant or of childbearing potential.
  * Known HIV seropositive, active hepatitis C infection, and/or hepatitis B (defined as HCV RNA

    ≥103 copies or HBV DNA ≥103 copies at screening).
  * Major surgical procedure within 28 days prior to the first dose of study treatment.
  * Presence of uncontrolled infection.
  * Evidence of active bleeding or bleeding diathesis.
  * Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | the duration from initiation of AraC treatment to the date of a first event or date of death from any cause, whichever come first, assessed up to 5 years
  Events were defined as a poor response to AraC, reactivation after AraC therapy and death from any cause.

SECONDARY OUTCOMES:
Overall response rate | on 12 months
  the cumulative number of patients with either non-active disease or regressive disease (signs and symptoms were improved with no new lesions) after AraC therapy
Overall survival | the duration from initiation of AraC treatment to the date of death or last follow-up, assessed up to 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, MD, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China